CLINICAL TRIAL: NCT04175496
Title: Glycemic and Insulinemic Responses of Low-Carbohydrate Snack Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zeynep Caferoglu, PhD, Assistant Professor Doctor, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ND
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: Glycemic index; Insulinemic index; Low carbohydrate; Snack; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Snacks; Cheese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Foods (Experimental): Blueberry Cake, Snack with Cheese and spicy Crackers will be used as test foods.
  Interventions: Other: Blueberry Cake; Other: Snacks with Cheese; Other: Spicy Crackers
- Reference Food (Experimental): Glucose solution will use as reference food.
  Interventions: Other: Glucose Solution First Repeat; Other: Glucose Solution Second Repeat

INTERVENTIONS:
Other: Blueberry Cake — Blueberry cake containing 25 g available CHO will be served to the participants after 10-hours fasting and asked to consume it within 15 minutes, along with 250 ml of water. Taking the first bite from test food will be considered as 0 min. Blood samples will be collected at time points 0,15, 30, 45, 60, 90 and 120 min.
  Arms: Test Foods
Other: Snacks with Cheese — Snacks with cheese containing 25 g available CHO will be served to the participants after 10-hours fasting and asked to consume it within 15 minutes, along with 250 ml of water. Taking the first bite from test food will be considered as 0 min. Blood samples will be collected at time points 0,15, 30, 45, 60, 90 and 120 min.
  Arms: Test Foods
Other: Spicy Crackers — Spicy crackers containing 25 g available CHO will be served to the participants after 10-hours fasting and asked to consume it within 15 minutes, along with 250 ml of water. Taking the first bite from test food will be considered as 0 min. Blood samples will be collected at time points 0,15, 30, 45, 60, 90 and 120 min.
  Arms: Test Foods
Other: Glucose Solution First Repeat — The glucose solution will be prepared by dissolving 25 g of glucose in 250 ml of water. Participants consume the glucose solution within 15 minutes after 10-hours fasting. Blood samples will be collect at time points 0,15, 30, 45, 60, 90 and 120 min.
  Arms: Reference Food
Other: Glucose Solution Second Repeat — The glucose solution will be prepared by dissolving 25 g of glucose in 250 ml of water. Participants consume the glucose solution within 15 minutes after 10-hours fasting. Blood samples will be collect at time points 0,15, 30, 45, 60, 90 and 120 min.
  Arms: Reference Food

SUMMARY:
The aim of this study is develop recipes containing CHO less than ICR, prepare new snacks alternatives that could be consumed without need for additional insulin doses, and evaluate the glycemic and insulinemic responses of these recipes. A randomized crossover trial will include 15 healthy adults aged 19-30 years. All participants will consume 3 test foods and reference food (glucose solution, 2 times) in a random order. Blood samples will be collected at time points 0,15, 30, 45, 60, 90 and 120 min. Glucose and insulin analyzes will be performed from blood samples. The results of these time points will be marked on the chart and the incremental area under the curve (iAUC) will be calculated for both glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Normal body weight (18.5-25 kg / m2 BMI)
* 19-30 years old

Exclusion Criteria:

* use of tobacco,
* weight change of >5 kg in the last 3 months
* the presence of any chronic disease or lactose intolerance,
* regular medicine use,
* pregnancy or lactation,
* performing competitive sports or endurance sports,
* fasting plasma glucose concentration >100 mg / dL,
* the presence of eating disorder,
* sensitivity or allergies to any food that used in the study

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose response | two hours postprandial period
  Postprandial glucose response will be quantified as incremental area under the curve (iAUC) (mg/dL x minutes), which is calculated according to the trapezoidal rule by using blood glucose values at time points 0, 15, 30, 45, 60, 90, and 120 minutes.
Postprandial insulin response | two hours postprandial period
  Postprandial insulin response will be quantified as incremental area under the curve (iAUC) (mg/dL x minutes), which is calculated according to the trapezoidal rule by using blood glucose values at time points 0, 15, 30, 45, 60, 90, and 120 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Health Sciences, Kayseri, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT04175496/Prot_SAP_000.pdf